CLINICAL TRIAL: NCT06574737
Title: Use of Surface Electromyography as a Tools to Predict Upper Extremity Recovery Function After Stroke
Status: Recruiting | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Other Study IDs: IKFR-202408.01
Record Dates: First submitted 2024-08-12; First posted 2024-08-28 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Upper Extremity Paresis; Muscle Contracture Upper Arm; Stroke
Keywords: Surface electromyography; Predictor Stroke; Upper Extremity Recovery
MeSH Terms: conditions — Paresis; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypothesis :

Based on the framework and premises above, the hypothesis is formulated as follows: H0 : surface electromyography parameters cannot predicts upper extremity motor function recovery in stroke patients H1: surface electromyography parameters can predicts upper extremity motor function recovery in stroke patients

DETAILED DESCRIPTION:
Study design and setting This study is an analytic quantitative observational study, to analyse the quantification of Manual Muscle Test score, Fugl Mayer Assessment-Upper Extremity score and electrical signals of the anterior deltoid, biceps, triceps, wrist flexors and wrist extensors muscles based on contractions, length of contraction and amplitude parameters in patients with acute phase stroke. This study performed at HasanSadikin Hospital between February 2024 - July 2024. Study participants Potential participants will be recruited by the main researcher

Inclusion criteria:

1. Patients who are hospitalized with upper extremity weakness due to stroke on the same side which confirmed with computed tomography scan or structural magnetic resonance imaging, in the acute phase
2. Men and women aged more than 18 years old
3. Willing to participate

Exclusion criteria:

1. Cognitive impairment (MoCA-Ina score less than 26)
2. Impaired consciousness (GCS score less than 15)
3. Unstable medical conditions at time of hospitalization
4. Patients with pacemaker
5. Having other injury or dysfunction in the impaired side of upper extremity that caused restrictions on the range of joint movement and muscle weakness, such as fractures, periarthritis, or moderate-severe pain
6. Diagnosis of other neurological disease or disorders in addition to stroke (e.g., traumatic brain injury, neuropathy or radiculopathy)
7. Get treated in isolation room
8. Hypersensitivity to gel electrodes

Drop out criteria:

1. Unable to do 2 or more follow up session
2. Withdrawn by themselves

Confounding factor:

1. Stroke location
2. Stroke size
3. Spasticity
4. Rehabilitation program
5. Compliance rehabilitation
6. Stroke risk factor

Sampling Technique The method of sampling based on consecutive samplings, that is, all stroke patients who meet the inclusion and exclusion criteria during the duration of the study.

Based on the formula above, the minimum sample size for this research is adequate, so the minimum sample size is 30 samples.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are hospitalized with upper extremity weakness due to stroke on the same side which confirmed with computed tomography (CT) scan or structural magnetic resonance imaging (MRI), in the acute phase
2. Men and women aged more than 18 years old
3. Willing to participate

Exclusion Criteria:

1. Cognitive impairment (MoCA-Ina score less than 26)
2. Impaired consciousness (GCS score less than 15)
3. Unstable medical conditions at time of hospitalization
4. Patients with pacemaker
5. Having other injury or dysfunction in the impaired side of upper extremity that caused restrictions on the range of joint movement and muscle weakness, such as fractures, periarthritis, or moderate-severe pain
6. Diagnosis of other neurological disease or disorders in addition to stroke (e.g., traumatic brain injury, neuropathy or radiculopathy)
7. Get treated in isolation room
8. Hypersensitivity to gel electrodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All stroke patients who meet the inclusion and exclusion criteria during the duration of the study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Electrical activity deltoid, biceps, triceps, wrist flexor, wrist extensor muscle | 3 days of stroke onset, 5 days of stroke onset, 1 months, 2 months and 3 months after stroke onset
  * Contraction (number/minute). The number of contractions was reported for each participant as a count of the number of contractions divided per minute time (the more the better outcome) windows analyzed for that participant.
  * Length of contraction (millisecond) (the longer the better outcome)
  * Amplitude (mV) (the more the better outcome)

SECONDARY OUTCOMES:
Manual Muscle Testing score | 3 days of stroke onset, 5 days of stroke onset, 1 months, 2 months and 3 months after stroke onset
  5: Normal 4: Good 3: Fair 2: Poor
  1: Trace 0: Zero
  (5 : higher end of strength ability, 0 = low-end ability of strength ability) (the more, the better outcome)
Fugl Mayer Assessment-Upper Extremity score | 3 days of stroke onset, 5 days of stroke onset, 1 months, 2 months and 3 months after stroke onset
  ≤25 : severe 26-45 : moderate 46-66 : mild
  (66 : maximum score for upper extremity score = normal, the more the better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Berthy Al Mungiza, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Sex Women Men Age Length of stay Stroke diagnosis Ischemic stroke Haemorrhagic stroke Stroke side Right hemisphere Left hemisphere Dominant Hand Right Left Stroke severity Minor stroke Moderate stroke Moderate to severe stroke Severe stroke Stroke risk factor Hypertension Diabetes Mellitus Heart disease Dyslipidemia Smoking Recurrent stroke Yes No
Supporting Information: Study Protocol, SAP
Time Frame: February 2025 - July 2025
Access Criteria: With access article/journal
  With participants characteristics:
  Sex Women Men Age Length of stay Stroke diagnosis Ischemic stroke Haemorrhagic stroke Stroke side Right hemisphere Left hemisphere Dominant Hand Right Left Stroke severity Minor stroke Moderate stroke Moderate to severe stroke Severe stroke Stroke risk factor Hypertension Diabetes Mellitus Heart disease Dyslipidemia Smoking Recurrent stroke Yes No

REFERENCES:
- [Result] Fan J, Li X, Yu X, Liu Z, Jiang Y, Fang Y, Zong M, Suo C, Man Q, Xiong L. Global Burden, Risk Factor Analysis, and Prediction Study of Ischemic Stroke, 1990-2030. Neurology. 2023 Jul 11;101(2):e137-e150. doi: 10.1212/WNL.0000000000207387. Epub 2023 May 17. PMID 37197995
- [Result] Venketasubramanian N, Yudiarto FL, Tugasworo D. Stroke Burden and Stroke Services in Indonesia. Cerebrovasc Dis Extra. 2022;12(1):53-57. doi: 10.1159/000524161. Epub 2022 Mar 21. PMID 35313314
- [Result] Shelton FN, Reding MJ. Effect of lesion location on upper limb motor recovery after stroke. Stroke. 2001 Jan;32(1):107-12. doi: 10.1161/01.str.32.1.107. PMID 11136923
- [Result] Lawrence ES, Coshall C, Dundas R, Stewart J, Rudd AG, Howard R, Wolfe CD. Estimates of the prevalence of acute stroke impairments and disability in a multiethnic population. Stroke. 2001 Jun;32(6):1279-84. doi: 10.1161/01.str.32.6.1279. PMID 11387487
- [Result] Feldner HA, Papazian C, Peters KM, Creutzfeldt CJ, Steele KM. Clinical Use of Surface Electromyography to Track Acute Upper Extremity Muscle Recovery after Stroke: A Descriptive Case Study of a Single Patient. Appl Syst Innov. 2021 Jun;4(2):32. doi: 10.3390/asi4020032. Epub 2021 May 10. PMID 34778722
- [Result] Steele KM, Papazian C, Feldner HA. Muscle Activity After Stroke: Perspectives on Deploying Surface Electromyography in Acute Care. Front Neurol. 2020 Sep 23;11:576757. doi: 10.3389/fneur.2020.576757. eCollection 2020. PMID 33071953
- [Result] Alt Murphy M, Al-Shallawi A, Sunnerhagen KS, Pandyan A. Early prediction of upper limb functioning after stroke using clinical bedside assessments: a prospective longitudinal study. Sci Rep. 2022 Dec 21;12(1):22053. doi: 10.1038/s41598-022-26585-1. PMID 36543863
- [Result] Papazian C, Baicoianu NA, Peters KM, Feldner HA, Steele KM. Electromyography Recordings Detect Muscle Activity Before Observable Contractions in Acute Stroke Care. Arch Rehabil Res Clin Transl. 2021 Jun 5;3(3):100136. doi: 10.1016/j.arrct.2021.100136. eCollection 2021 Sep. PMID 34589686
- [Result] Stinear CM, Smith MC, Byblow WD. Prediction Tools for Stroke Rehabilitation. Stroke. 2019 Nov;50(11):3314-3322. doi: 10.1161/STROKEAHA.119.025696. Epub 2019 Oct 15. No abstract available. PMID 31610763
- [Result] Manzur-Valdivia H, Alvarez-Ruf J. Surface Electromyography in Clinical Practice. A Perspective From a Developing Country. Front Neurol. 2020 Oct 15;11:578829. doi: 10.3389/fneur.2020.578829. eCollection 2020. PMID 33178121
- [Result] Ueda S, Aoki H, Yasuda Y, Nishiyama A, Hayashi Y, Honaga K, Tanuma A, Takakura T, Kurosu A, Hatori K, Hayashi A, Fujiwara T. The MMT of Elbow Flexion and the AFE Predict Impairment and Disability at 3 Weeks in Patients With Acute Stroke. Front Neurol. 2022 Mar 30;13:831800. doi: 10.3389/fneur.2022.831800. eCollection 2022. PMID 35432154
- [Result] Lv W, Liu K, Zhou P, Huang F, Lu Z. Surface EMG analysis of weakness distribution in upper limb muscles post-stroke. Front Neurol. 2023 Apr 25;14:1135564. doi: 10.3389/fneur.2023.1135564. eCollection 2023. PMID 37181551
- [Result] Raghavan P. Upper Limb Motor Impairment After Stroke. Phys Med Rehabil Clin N Am. 2015 Nov;26(4):599-610. doi: 10.1016/j.pmr.2015.06.008. Epub 2015 Aug 25. PMID 26522900
- [Result] Li S. Stroke Recovery Is a Journey: Prediction and Potentials of Motor Recovery after a Stroke from a Practical Perspective. Life (Basel). 2023 Oct 15;13(10):2061. doi: 10.3390/life13102061. PMID 37895442
- [Result] Grefkes C, Fink GR. Recovery from stroke: current concepts and future perspectives. Neurol Res Pract. 2020 Jun 16;2:17. doi: 10.1186/s42466-020-00060-6. eCollection 2020. PMID 33324923
- [Result] Pregnolato G, Rimini D, Baldan F, Maistrello L, Salvalaggio S, Celadon N, Ariano P, Pirri CF, Turolla A. Clinical Features to Predict the Use of a sEMG Wearable Device (REMO(R)) for Hand Motor Training of Stroke Patients: A Cross-Sectional Cohort Study. Int J Environ Res Public Health. 2023 Mar 14;20(6):5082. doi: 10.3390/ijerph20065082. PMID 36981992
- [Result] Salvalaggio S, Boccuni L, Turolla A. Patient's assessment and prediction of recovery after stroke: a roadmap for clinicians. Arch Physiother. 2023 Jun 19;13(1):13. doi: 10.1186/s40945-023-00167-4. PMID 37337288
- [Result] Roman NA, Miclaus RS, Nicolau C, Sechel G. Customized Manual Muscle Testing for Post-Stroke Upper Extremity Assessment. Brain Sci. 2022 Mar 28;12(4):457. doi: 10.3390/brainsci12040457. PMID 35447988
- [Result] Kostka J, Niwald M, Guligowska A, Kostka T, Miller E. Muscle power, contraction velocity and functional performance after stroke. Brain Behav. 2019 Apr;9(4):e01243. doi: 10.1002/brb3.1243. Epub 2019 Feb 28. PMID 30821102
- [Result] Pandian S, Arya KN. Stroke-related motor outcome measures: do they quantify the neurophysiological aspects of upper extremity recovery? J Bodyw Mov Ther. 2014 Jul;18(3):412-23. doi: 10.1016/j.jbmt.2013.11.006. Epub 2013 Nov 9. PMID 25042312
- [Result] McManus L, De Vito G, Lowery MM. Analysis and Biophysics of Surface EMG for Physiotherapists and Kinesiologists: Toward a Common Language With Rehabilitation Engineers. Front Neurol. 2020 Oct 15;11:576729. doi: 10.3389/fneur.2020.576729. eCollection 2020. PMID 33178118
- [Result] Hogrel JY. Clinical applications of surface electromyography in neuromuscular disorders. Neurophysiol Clin. 2005 Jul;35(2-3):59-71. doi: 10.1016/j.neucli.2005.03.001. PMID 16087069

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT06574737/Prot_SAP_ICF_000.pdf